CLINICAL TRIAL: NCT07189637
Title: The Combined Effect of the Mediterranean Diet and Intermittent Fasting on Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nadide Gizem Tarakci Filiz (Other)
Collaborators: Medipol University (Other); Istanbul Medipol University Hospital (Other); Fenerbahce University (Other)
Responsible Party: Sponsor-Investigator, Nadide Gizem Tarakci Filiz, Asst. Prof., Fenerbahce University
Organization: Fenerbahce University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-3317; 2025/48 (Other Grant/Funding Number: Istanbul Medipol University)
Record Dates: First submitted 2025-09-13; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: Hypertension; Cardiovascular diseases; DASH diet; Mediterranean diet; Intermittent fasting
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Intermittent Fasting | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (control) (Other): Participants will only receive face-to-face nutrition education.
  Interventions: Other: Face-to-face nutrition education
- Group B (Intermittent Fasting Diet Group) (Experimental): Participants will receive face-to-face nutrition education and Intermittent Fasting Diet. Additionally, a brochure package containing information about Intermittent Fasting Diet models will be prepared by a dietitian and distributed to participants by the same dietitian along with the training.
  Interventions: Other: Face-to-face nutrition education; Other: Intermittent Fasting Diet
- Group C (Mediterranean Diet Group) (Experimental): Participants will receive face-to-face nutrition education and Mediterranean Diet. Additionally, a brochure package containing information about Mediterranean Diet models will be prepared by a dietitian and distributed to participants by the same dietitian along with the training.
  Three separate packages compliant with the Mediterranean Diet will be given at the start of the study, 2nd week and 4th week.
  Package 1: 250 mL natural extra virgin olive oil, 150 g walnuts, 1 avocado, 250 g black raisins, 1 L semi-skimmed UHT cow's milk, 1 kg green lentils and 1 garlic clove Package 2: 250 mL of natural extra virgin olive oil, 200 g of raw hazelnuts, 150-200 g of unsalted black olives, 140 g of dried apricots, 1 L of semi-skimmed UHT cow's milk, 1 kg of dried beans, and 700 g of unsalted tomato paste Package 3: 250 mL extra virgin olive oil, 180 g unsalted pumpkin seeds, 1 kg apples, 1 L semi-skimmed UHT cow's milk, 500 g whole wheat pasta and 500 g red lentils
  Interventions: Other: Face-to-face nutrition education; Other: Mediterranean Diet
- Group D (the Combination of Intermittent Fasting Diet and Mediterranean Diet) (Experimental): Participants will receive face-to-face nutrition education and the combination of IFD and MD. Additionally, a brochure package containing information about IFD and MD models will be prepared by a dietitian and distributed to participants by the same dietitian along with the training.
  Three separate packages compliant with the MD will be given at the start of the study, 2nd week and 4th week.
  Pkg. 1: 250 mL natural extra virgin olive oil, 150 g walnuts, 1 avocado, 250 g black raisins, 1 L semi-skimmed UHT cow's milk, 1 kg green lentils and 1 garlic clove Pkg. 2: 250 mL of natural extra virgin olive oil, 200 g of raw hazelnuts, 150-200 g of unsalted black olives, 140 g of dried apricots, 1 L of semi-skimmed UHT cow's milk, 1 kg of dried beans, and 700 g of unsalted tomato paste Pkg. 3: 250 mL extra virgin olive oil, 180 g unsalted pumpkin seeds, 1 kg apples, 1 L semi-skimmed UHT cow's milk, 500 g whole wheat pasta and 500 g red lentils
  Interventions: Other: Face-to-face nutrition education; Other: Intermittent Fasting Diet; Other: Mediterranean Diet

INTERVENTIONS:
Other: Face-to-face nutrition education — All participants will receive face-to-face nutrition education from specialist dietitians in accordance with the principles of nutrition for hypertension. Nutrition education will be provided through prepared brochures. The brochures will be given to participants as gifts. Nutrition education will cover topics such as hypertension and nutrition, nutrients, the importance of micronutrients, foods containing salt, reading labels, limiting salt consumption, healthy fat consumption, fibre consumption, water consumption, and healthy cooking methods.
Other: Intermittent Fasting Diet — Training will be provided to all participants through a food and nutrition photo catalogue so that portions can be recorded correctly and within standard limits when keeping a food diary. Participants will restrict their food intake to a 16-hour period by applying the 16/8 Intermittent Fasting Diet model and will eat and drink whatever they want during the remaining 8 hours. During this 16-hour period, they will consume non-energy drinks consisting of water, unsweetened tea, unsweetened herbal teas and black coffee. It will be recommended that intermittent fasting be maintained from 6:00 p.m. to 10:00 a.m. However, participants may also choose other 16-hour periods, such as 7:00 p.m. to 11:00 a.m. or 8:00 p.m. to 12:00 p.m. Participants will be given a tracking chart to record the first and last times they consume food or energy-containing beverages during the day, and their adherence to the diet will be monitored based on their declarations.
  Arms: Group B (Intermittent Fasting Diet Group); Group D (the Combination of Intermittent Fasting Diet and Mediterranean Diet)
Other: Mediterranean Diet — Training will be provided to all participants through a food and nutrition photo catalogue to ensure that portions are recorded correctly and within standard limits when keeping a food diary. In addition, the dietician will provide this group with a diet plan calculated for energy, macro and micro nutrients, which will be different each week for the first four follow-ups. The diet plans provided will be prepared in accordance with the Mediterranean Diet food pyramid. Participants' energy requirements will be calculated using the Schofield Equation for basal metabolic rate, with adjustments made according to their physical activity levels. Energy requirements will be met by 45-50% from carbohydrates, 15-20% from protein, and 25-35% from fats.
  Arms: Group C (Mediterranean Diet Group); Group D (the Combination of Intermittent Fasting Diet and Mediterranean Diet)

SUMMARY:
Hypertension (HT) is an important risk factor for cardiovascular diseases (CVD) and death. Approximately 16.9 million people in Turkey have HT. Nutritional habits play an important role in the development of HT. DASH (Dietary Approaches to Stop Hypertension) and the Mediterranean diet (MD) have been found to be effective in lowering blood pressure and reducing cardiometabolic risks. The DASH diet stands out with its low sodium, saturated fat, simple sugar and cholesterol content, while it is rich in fiber, potassium, magnesium and anti-inflammatory components. The MD is based on healthy foods such as olive oil, vegetables, fruits, fish and nuts, and contains antioxidants and healthy fatty acids. This study will investigate whether the sodium-restricted MD can offer a model comparable to DASH. In addition, the effects of the intermittent fasting diet (IFD) model alone and in combination with the MD on blood pressure will be examined. It has been observed that IFD reduces blood pressure by reducing energy intake and acting on the autonomic nervous system. The aim of this project is to evaluate the effects of MD, IFD and both of them on hypertension and to present a new and original approach in this field.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed hypertension patients
* Individuals with blood pressure >140/90 mmHg
* Individuals with a body mass index (BMI) in the range of 18.5-25 kg/m²
* Individuals aged 40-65 years

Exclusion Criteria:

Participants will be excluded if they have any of the following:

* Type 2 Diabetes Mellitus
* Type 1 Diabetes Mellitus
* Cardiovascular disease
* Liver disease
* Kidney disease
* Gastrointestinal disease
* Respiratory disease
* Psychiatric disorders
* Women who are pregnant or breastfeeding
* Severe food allergies
* Current smokers or individuals consuming alcohol regularly
* History of major surgery within the last 6 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | At enrollment, 1 week later than enrollment, 2 weeks later than enrollment, 3 weeks later than enrollment, 4 weeks later than enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  The participants' blood pressure will be measured six times in this research. Blood pressure measurements will be taken by a trained physician in accordance with standard measurement protocols. Measurements will be taken after a 5-minute rest period, with the patient seated, using an automatic blood pressure monitor with the correct cuff size applied to the arm. Two consecutive measurements will be taken for each patient, with at least 1 minute between measurements. The average of the two measurements obtained will be used in the analyses.
  The following points will be taken into consideration during the measurements.
  * Patients should not have smoked, consumed caffeine, or exercised in the last 30 minutes
  * During the measurement, the patient should be leaning back with their feet flat on the floor
  * The arm being measured should be supported at heart level Blood pressure values will be evaluated according to the 2023 ESC/ESH hypertension guidelines.

SECONDARY OUTCOMES:
Height in cm | At enrollment, 1 week later than enrollment, 2 weeks later than enrollment, 3 weeks later than enrollment, 4 weeks later than enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  Height measurement will be taken by a specialist dietician. It will be performed in accordance with the measurement techniques and standards recommended by the International Society for the Advancement of Kinanthropometry. Participants' heights will be measured barefoot using a stadiometer with an accuracy of 0.01 m.
Body weight in kg | At enrollment, 1 week later than enrollment, 2 weeks later than enrollment, 3 weeks later than enrollment, 4 weeks later than enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  Body weight measurement will be taken by a specialist dietician. It will be performed in accordance with the measurement techniques and standards recommended by the International Society for the Advancement of Kinanthropometry. Body weight and body composition will be measured using a body composition analyser with a precision of 0.1 kg. The participants' clothing weight (1.0 kg) will be recorded on the analyser before measurement. Measurements will be taken barefoot and with participants wearing light clothing. Metal objects on participants will be removed.
Body Mass Index (BMI) in kg/m² | At enrollment, 1 week later than enrollment, 2 weeks later than enrollment, 3 weeks later than enrollment, 4 weeks later than enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  Body Mass Index (BMI) will be used to assess whether an individual's body weight is appropriate for their height. It is calculated by dividing a person's body weight, measured in kilograms (kg), by the square of their height, measured in meters (m). Since height will be measured in centimeters (cm), it will first be converted into meters. This will be done by dividing the height in centimeters by 100.
Waist circumference in cm | At enrollment, 1 week later than enrollment, 2 weeks later than enrollment, 3 weeks later than enrollment, 4 weeks later than enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  Waist circumference: Waist circumference will be taken by a specialist dietician. It will be measured at the narrowest point of the waist with the individual standing upright and without any clothing around the waist. Measurements will be taken with a tape measure, ensuring it is in contact with the skin without applying excessive pressure.
Fasting plasma glucose in mg/dL | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: 70-99 mg/dL
HbA1c in % | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: < 5.7% (normal), 5.7-6.4% (prediabetes), ≥ 6.5% (diabetes)
Insulin in µU/mL | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: 2-25 µU/mL
Triglycerides in mg/dL | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: < 150 mg/dL
HDL cholesterol in mg/dL | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values:
  Men: ≥ 40 mg/dL Women: ≥ 50 mg/dL
LDL cholesterol in mg/dL | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: < 100 mg/dL
Total cholesterol in mg/dL | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: < 200 mg/dL
Urea in mg/dL | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: 7-20 mg/dL
Creatinine in mg/dL | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values:
  Men: 0.7-1.3 mg/dL Women: 0.6-1.1 mg/dL
Sodium in mmol/L | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: 135-145 mmol/L
Potassium in mmol/L | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: 3.5-5.0 mmol/L
hs-CRP in mg/L | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: < 1 mg/L (low cardiovascular risk), 1-3 mg/L (intermediate risk), > 3 mg/L (high risk)
ALT in U/L | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: Men: < 41 U/L; Women: < 31 U/L
AST in U/L | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: Men: < 40 U/L; Women: < 32 U/L
GGT in U/L | At enrollment, 13 weeks later than enrollment, 26 weeks later than enrollment
  This will be obtained from blood tests. Reference values: Men: 8-61 U/L; Women: 5-36 U/L

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet KOÇAK, PhD, Principal Investigator — İstanbul Medipol Üniversitesi/Sağlık Bilim Ve Teknolojileri Araştırma Enstitüsü
Locations (1):
- Medipol Mega University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Filippou C, Thomopoulos C, Konstantinidis D, Siafi E, Tatakis F, Manta E, Drogkaris S, Polyzos D, Kyriazopoulos K, Grigoriou K, Tousoulis D, Tsioufis K. DASH vs. Mediterranean diet on a salt restriction background in adults with high normal blood pressure or grade 1 hypertension: A randomized controlled trial. Clin Nutr. 2023 Oct;42(10):1807-1816. doi: 10.1016/j.clnu.2023.08.011. Epub 2023 Aug 18. PMID 37625311
- [Background] Zou Y, Tang J, Zhang F, Chen D, Mu L, Xu H, Yu P, Ren Y, Mei Y, Mu L. Effect of low-sodium salt applied to Chinese modified DASH diet on arterial stiffness in older patients with hypertension and type 2 diabetes. Nutr Hosp. 2023 Oct 6;40(5):967-974. doi: 10.20960/nh.04622. PMID 37534516
- [Background] Zhou X, Lin X, Yu J, Yang Y, Muzammel H, Amissi S, Schini-Kerth VB, Lei X, Jose PA, Yang J, Shi D. Effects of DASH diet with or without time-restricted eating in the management of stage 1 primary hypertension: a randomized controlled trial. Nutr J. 2024 Jun 17;23(1):65. doi: 10.1186/s12937-024-00967-9. PMID 38886740
- [Background] Zhou B, Perel P, Mensah GA, Ezzati M. Global epidemiology, health burden and effective interventions for elevated blood pressure and hypertension. Nat Rev Cardiol. 2021 Nov;18(11):785-802. doi: 10.1038/s41569-021-00559-8. Epub 2021 May 28. PMID 34050340
- [Background] Guideline: Sodium Intake for Adults and Children. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK133309/ PMID 23658998
- [Background] World Health Organization (WHO). "Obesity and overweight". https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight. Last access: 12.02.2024
- [Background] Valenzuela-Fuenzalida JJ, Bravo VS, Valarezo LM, Delgado Retamal MF, Leiva JM, Bruna-Mejias A, Nova-Baeza P, Orellana-Donoso M, Suazo-Santibanez A, Oyanedel-Amaro G, Gutierrez-Espinoza H. Effectiveness of DASH Diet versus Other Diet Modalities in Patients with Metabolic Syndrome: A Systematic Review and Meta-Analysis. Nutrients. 2024 Sep 10;16(18):3054. doi: 10.3390/nu16183054. PMID 39339654
- [Background] Urquiaga I, Echeverria G, Dussaillant C, Rigotti A. [Origin, components and mechanisms of action of the Mediterranean diet]. Rev Med Chil. 2017 Jan;145(1):85-95. doi: 10.4067/S0034-98872017000100012. Spanish. PMID 28393974
- [Background] The International Society for the Advancement of Kinanthropometry. www.isak.global. Last access: 03.11.2023
- [Background] Stekovic S, Hofer SJ, Tripolt N, Aon MA, Royer P, Pein L, Stadler JT, Pendl T, Prietl B, Url J, Schroeder S, Tadic J, Eisenberg T, Magnes C, Stumpe M, Zuegner E, Bordag N, Riedl R, Schmidt A, Kolesnik E, Verheyen N, Springer A, Madl T, Sinner F, de Cabo R, Kroemer G, Obermayer-Pietsch B, Dengjel J, Sourij H, Pieber TR, Madeo F. Alternate Day Fasting Improves Physiological and Molecular Markers of Aging in Healthy, Non-obese Humans. Cell Metab. 2019 Sep 3;30(3):462-476.e6. doi: 10.1016/j.cmet.2019.07.016. Epub 2019 Aug 27. PMID 31471173
- [Background] McClave SA, Martindale RG, Vanek VW, McCarthy M, Roberts P, Taylor B, Ochoa JB, Napolitano L, Cresci G; A.S.P.E.N. Board of Directors; American College of Critical Care Medicine; Society of Critical Care Medicine. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2009 May-Jun;33(3):277-316. doi: 10.1177/0148607109335234. No abstract available. PMID 19398613
- [Background] Schwingshackl L, Hoffmann G. Mediterranean dietary pattern, inflammation and endothelial function: a systematic review and meta-analysis of intervention trials. Nutr Metab Cardiovasc Dis. 2014 Sep;24(9):929-39. doi: 10.1016/j.numecd.2014.03.003. Epub 2014 Apr 2. PMID 24787907
- [Background] Schofield WN. Predicting basal metabolic rate, new standards and review of previous work. Hum Nutr Clin Nutr. 1985;39 Suppl 1:5-41. PMID 4044297
- [Background] Saulle, R., La Torre, G. 2010. "The Mediterranean Diet, recognized by UNESCO as a cultural heritage of humanity", Italian Journal of Public Health, 7(4).
- [Background] Sacks FM, Campos H. Dietary therapy in hypertension. N Engl J Med. 2010 Jun 3;362(22):2102-12. doi: 10.1056/NEJMct0911013. No abstract available. PMID 20519681
- [Background] Raymond, J. L., Morrow, K. 2021. "Dietary Approaches to Stop Hypertension (DASH) Diet". Appendix 17. In: Krause and Mahan's Food and the Nutrition Care Process. Elsevier. 15 th Edition ISBN Number: 978-0-323-63655-1, 1047-1048.
- [Background] Rakıcıoğlu, N., Acar Tek, N., Ayaz, A., Pekcan, G. 2009. "Food and Nutrition Photo Catalogue". 2nd edition. Ata Ofset Yayın Evi. Ankara.
- [Background] Pehlivanoğlu, E. F. Ö., Balcioğlu, H., Ünlüoğlu, İ. 2020. "Validity and reliability of adapting the Mediterranean diet adherence scale into Turkish", Osmangazi Medical Journal, 42(2), 160-164.
- [Background] Park YM, Steck SE, Fung TT, Zhang J, Hazlett LJ, Han K, Lee SH, Kwon HS, Merchant AT. Mediterranean diet, Dietary Approaches to Stop Hypertension (DASH) style diet, and metabolic health in U.S. adults. Clin Nutr. 2017 Oct;36(5):1301-1309. doi: 10.1016/j.clnu.2016.08.018. Epub 2016 Sep 8. PMID 27665232
- [Background] National Institutes of Health. 2020. "Addressing the inclusion of older adults in clinical trials (NIH Publication No. 20-12345)". U.S. Department of Health and Human Services. https://www.nih.gov/sites/default/files/publications/20-12345.pdf. Last access: 10.01.2024.
- [Background] Martin, R. 1957. "Lehrbuch der antropologie". Saller, K. (Ed.). (3th ed.). Stuttgart: G. Fisher Verlag
- [Background] Marfell-Jones, M., Olds, T., Stewart, A., Stewart-Oaten, A., Jones, M., Ridder, W. H. 2001. "International Society for the Advancement of Kinanthropometry". International standards for anthropometric assessment.
- [Background] Malinowski B, Zalewska K, Wesierska A, Sokolowska MM, Socha M, Liczner G, Pawlak-Osinska K, Wicinski M. Intermittent Fasting in Cardiovascular Disorders-An Overview. Nutrients. 2019 Mar 20;11(3):673. doi: 10.3390/nu11030673. PMID 30897855
- [Background] Magriplis E, Panagiotakos D, Kyrou I, Tsioufis C, Mitsopoulou AV, Karageorgou D, Dimakopoulos I, Bakogianni I, Chourdakis M, Micha R, Michas G, Ntouroupi T, Tsaniklidou SM, Argyri K, Zampelas A. Presence of Hypertension Is Reduced by Mediterranean Diet Adherence in All Individuals with a More Pronounced Effect in the Obese: The Hellenic National Nutrition and Health Survey (HNNHS). Nutrients. 2020 Mar 23;12(3):853. doi: 10.3390/nu12030853. PMID 32209978
- [Background] Lv Y, Aihemaiti G, Guo H. Effect of Dietary Approaches to Stop Hypertension (DASH) on Patients with Metabolic Syndrome and Its Potential Mechanisms. Diabetes Metab Syndr Obes. 2024 Aug 23;17:3103-3110. doi: 10.2147/DMSO.S477739. eCollection 2024. PMID 39206416
- [Background] Lim CY, In J. Randomization in clinical studies. Korean J Anesthesiol. 2019 Jun;72(3):221-232. doi: 10.4097/kja.19049. Epub 2019 Apr 1. PMID 30929415
- [Background] Keys A. Mediterranean diet and public health: personal reflections. Am J Clin Nutr. 1995 Jun;61(6 Suppl):1321S-1323S. doi: 10.1093/ajcn/61.6.1321S. PMID 7754982
- [Background] Hipertansiyon Tani ve Tedavi Kılavuzu. Türkiye Endokrinoloji ve Metabolizma Derneği. 2022 ISBN: 978-605-66410-4-6
- [Background] Gonzalez JE, Cooke WH. Influence of an acute fast on ambulatory blood pressure and autonomic cardiovascular control. Am J Physiol Regul Integr Comp Physiol. 2022 Jun 1;322(6):R542-R550. doi: 10.1152/ajpregu.00283.2021. Epub 2022 Apr 5. PMID 35380473
- [Background] Filippou C, Tatakis F, Polyzos D, Manta E, Thomopoulos C, Nihoyannopoulos P, Tousoulis D, Tsioufis K. Overview of salt restriction in the Dietary Approaches to Stop Hypertension (DASH) and the Mediterranean diet for blood pressure reduction. Rev Cardiovasc Med. 2022 Jan 19;23(1):36. doi: 10.31083/j.rcm2301036. PMID 35092228
- [Background] Estruch, R., Ros E., Salas-Salvadó J., Covas, M. I., Corella, D., Arós, F., Gómez-Gracia, E., Ruiz-Gutiérrez, V., Fiol, M., Lapetra, J., Lamuela-Raventos, R. M., Serra-Majem, L., Pintó, X., Basora, J., Muñoz, M. A., Sorlí, J. V., Martínez, J. A., Fitó, M., Gea, A., Hernán, M. A., Martínez-González, M. A. 2018. "PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts", N Engl J Med, 21;378(25), 34.
- [Background] Erdem Y, Ozkan G, Ulusoy S, Arici M, Derici U, Sengul S, Sindel S, Erturk S; Turkish Society of Hypertension and Renal Diseases. The effect of intermittent fasting on blood pressure variability in patients with newly diagnosed hypertension or prehypertension. J Am Soc Hypertens. 2018 Jan;12(1):42-49. doi: 10.1016/j.jash.2017.11.008. Epub 2017 Dec 6. PMID 29275920
- [Background] Erdem NZ, Bayraktaroglu E, Samanci RA, Gecgil-Demir E, Tarakci NG, Mert-Biberoglu F. The effect of intermittent fasting diets on body weight and composition. Clin Nutr ESPEN. 2022 Oct;51:207-214. doi: 10.1016/j.clnesp.2022.08.030. Epub 2022 Aug 28. PMID 36184206
- [Background] Ebispro for Windows 8.0.Entwickelt an der Universitat Hohenheim; Stuttgart, Germany, 2012. Turkish Version (BEBIS), Pacific Electric Electronics. www.bebis. com.tr; Istanbul.
- [Background] de Cabo R, Mattson MP. Effects of Intermittent Fasting on Health, Aging, and Disease. N Engl J Med. 2019 Dec 26;381(26):2541-2551. doi: 10.1056/NEJMra1905136. No abstract available. PMID 31881139
- [Background] D'Alessandro A, De Pergola G. The Mediterranean Diet: its definition and evaluation of a priori dietary indexes in primary cardiovascular prevention. Int J Food Sci Nutr. 2018 Sep;69(6):647-659. doi: 10.1080/09637486.2017.1417978. Epub 2018 Jan 18. PMID 29347867
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Background] Barbaresko J, Koch M, Schulze MB, Nothlings U. Dietary pattern analysis and biomarkers of low-grade inflammation: a systematic literature review. Nutr Rev. 2013 Aug;71(8):511-27. doi: 10.1111/nure.12035. Epub 2013 Jun 13. PMID 23865797
- [Background] Anton SD, Moehl K, Donahoo WT, Marosi K, Lee SA, Mainous AG 3rd, Leeuwenburgh C, Mattson MP. Flipping the Metabolic Switch: Understanding and Applying the Health Benefits of Fasting. Obesity (Silver Spring). 2018 Feb;26(2):254-268. doi: 10.1002/oby.22065. Epub 2017 Oct 31. PMID 29086496
- [Background] Akbulut, G. 2017. "Current Mediterranean diet and potential health effects", Türkiye Clinics Journal of Health Sciences, 2(2).